CLINICAL TRIAL: NCT03613701
Title: Relationship Between Endothelial Progenitor Cells and Revascularization Effect of Moyamoya Disease
Acronym: REPCREMMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 8157113
Record Dates: First submitted 2018-07-29; First posted 2018-08-03 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Moyamoya Disease
Keywords: Moyamoya disease; Endothelial progenitor cells; revascularization
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moyamoya disease patients: Moyamoya disease patients/Healthy volunteers

SUMMARY:
Moyamoya disease is a chronic cerebrovascular disease，The typical pathological manifestations are the stenosis or occlusion of the distal internal carotid artery and/or middle cerebral artery, and the proximal anterior cerebral artery. Meanwhile, the abnormal vascular net, which is the smokey vessel, occurs at the bottom of the brain. Currently the pathogenesis of this disease is unknown. Limited studies have reported the expression of endothelial progenitor cells (EPCs) in moyamoya disease, but the results were inconsistent. Some investigators believe that the number of EPCs in peripheral blood of patients with moyamoya disease is increased, while others believe that the number of EPCs in peripheral blood of moyamoya patients is reduced. Therefore, the investigators need to find a more accurate detection method to confirm the growth of EPC in patients with moyamoya disease. At the same time, whether there is endothelial injury in patients with smoke disease, and the expression of endothelial cells (CEC) in patients with smoke disease, there is no research on this aspect at home and abroad.

DETAILED DESCRIPTION:
Objective: Detect the expression of endothelial progenitor cells and endothelial cells from peripheral blood of patients with moyamoya disease, and to assess the relationship between clinical characteristics.

Design: A single center study, and planned to enroll 120 patients. The present study was to detect the quantities of EPC from peripheral blood in Moyamoya disease by flow cytometry, and to identify the relationship of endothelial progeIlitor cells and effect of the revascularization on Moyamoya disease. The present study also use cerebral ischemia animal model foe intervention experiment, to explore whether EPC can promote vascular remodeling effect of ischemic cerebrovascular disease, and to provide new thought for the treatment of chronic cerebrovascular disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Whole-brain vessels angiography or magnetic resonance arteriography (MRA) has the following manifestations: stenosis or occlusion of terminal internal carotid artery or the anterior cerebral artery and/or initiating middle cerebral artery; In the arterial phase, the abnormal smokey vascular net near the occlusive or stenosis lesion can be seen.
2. For patients with stable stroke, there was no acute or subacute cerebral infarction or cerebral hemorrhage, and at least 3 months before the last cerebral infarction or cerebral hemorrhage events.

Exclusion Criteria:

1. Exclude atherosclerosis, autoimmune diseases, meningitis, intracranial tumors, multiple neurofibromatosis, Down syndrome, craniocerebral trauma, radiation injury, and other underlying diseases that may cause smoke.
2. Acute or subacute cerebral infarction or cerebral hemorrhage were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Health volunteers' inclusion criteria:
  1. Age between 18-60;
  2. Male or female;
  Exclusion criteria:
  Exclude the volunteers with history of cerebrovascular disease and heart disease.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Expression of endothelial progenitor cells and endothelial cells in peripheral blood | 2017.9-2018.8
  Expression of endothelial progenitor cells and endothelial cells in peripheral

CONTACTS AND LOCATIONS:
Overall Officials: Lian Duan, Chief, Study Chair — The 307th Hospital of Military Chinese People's Liberation Army
Locations (1):
- The 307th Hospital of Military Chinese People's Liberation Army, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao G, Liu SM, Hao FB, Wang MJ, Wang QN, Yang RM, Guo QB, Wang XP, Li JJ, Han C, Duan L, Zhang JN. Treatment for moyamoya disease with hyperhomocysteinemia. J Cereb Blood Flow Metab. 2025 Aug;45(8):1469-1478. doi: 10.1177/0271678X251325676. Epub 2025 Mar 13. PMID 40079509
- [Derived] Gao G, Hao FB, Wang QN, Wang XP, Liu SM, Wang MJ, Guo QB, Li JJ, Bao XY, Han C, Duan L. Surgical outcomes following encephaloduroarteriosynangiosis in moyamoya disease associated with hyperhomocysteinemia. Brain Behav. 2023 Aug;13(8):e3093. doi: 10.1002/brb3.3093. Epub 2023 Jun 29. PMID 37386744